CLINICAL TRIAL: NCT06293807
Title: Immediate Post-Operative Anesthesia With Either Lidocaine or Bupivacaine: A Short-term Clinical Response
Brief Title: Immediate Post-Operative Anesthesia With Either Lidocaine or Bupivacaine
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20220162HU
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Periodontal Diseases
Keywords: Flap debridement; Flap osseous; Tooth extractions; Guided Tissue Regeneration; IV sedation; Local anesthesia
MeSH Terms: conditions — Periodontal Diseases | interventions — Lidocaine; Epinephrine; Bupivacaine; Saline Solution

STUDY DESIGN:
Intervention Model Description: A randomized, placebo-controlled, parallel design study.
Who Masked: Participant, Investigator
Masking Description: Both the surgeon and patient will be blinded as to the intervention provided by covering identifying marks of the anesthetic carpules to be administered. Randomization will be assured by random selection of a slip of paper drawn from a sealed envelope assigning the patient to one of three groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment group Xylocaine (Experimental): Participants have been scheduled to receive an area of gum surgery to treat periodontal (gum) disease in their mouth while under intravenous (IV) conscious sedation. The study drug is administered after surgery.
  Interventions: Drug: Xylocaine 2 % with 1:100,000 epinephrine
- Treatment group Bupivicaine (Experimental): Participants have been scheduled to receive an area of gum surgery to treat periodontal (gum) disease in their mouth while under intravenous (IV) conscious sedation. The study drug is administered after surgery.
  Interventions: Drug: Bupivicaine 0.5% with 1:200,000 epinephrine
- Placebo control group (Placebo Comparator): Participants have been scheduled to receive an area of gum surgery to treat periodontal (gum) disease in their mouth while under intravenous (IV) conscious sedation. The study drug is administered after surgery.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Xylocaine 2 % with 1:100,000 epinephrine — Local anesthetic used during dental procedures
  Other Names: Lidocaine
  Arms: Treatment group Xylocaine
Drug: Bupivicaine 0.5% with 1:200,000 epinephrine — Local anesthetic used during dental procedures
  Other Names: Marcaine
  Arms: Treatment group Bupivicaine
Other: Placebo — 0.9% Normal Saline solution used in place of local anesthetic
  Other Names: Normal Saline 0.9%
  Arms: Placebo control group

SUMMARY:
Immediate post-suturing administration of either one of two dental anesthetic solutions or a placebo prior to dismissal.

DETAILED DESCRIPTION:
This study seeks to evaluate the pain response following the administration of two anesthetic solutions just prior to patient dismissal from a surgical procedure: 2% Xylocaine with 1:100,000 epi and 0.5% Bupivicaine with 1:200,000 epi in comparison with 0.9% Normal Saline as a placebo. the study team will monitor pain response following these interventions at 4, 8, 12, 24, and 48 hours.

ELIGIBILITY:
Inclusion Criteria:

-Patients who have undergone a comprehensive periodontal evaluation and treatment plan not related to participation in this study and…

1. require flap surgery of 2 to 5 teeth in a continuous site (including flap debridement, flap osseous, extractions, and Guided Tissue Regeneration (GTR) procedures), and…
2. require IV sedation and local anesthesia or local anesthesia only…
3. in either the maxillary or mandibular arch.

Exclusion Criteria:

1. Pregnancy, or those planning to become pregnant
2. allergy or any medical issue using Lidocaine or Bupivacaine
3. inability to take non-steroidal anti-inflammatory drugs (NSAIDS) or acetaminophen
4. non-English speaking
5. not possessing an I-phone or Android device
6. patients requiring narcotic for IV sedation
7. patients requiring either IV or oral steroids during the perioperative period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2023-04-16 (Actual); Study Completion 2023-04-16 (Actual)

PRIMARY OUTCOMES:
Change in pain using Visual Analog Scale (VAS) | Baseline to 48 hours
  Pain response recorded using a 20 point visual Analog Scale. The VAS scale is a straight line scale scored from 0-20 with 0 indicating the least amount of pain and 20 the worst pain ever experienced.
Number of Ibuprofen administered | Baseline to 48 hours
  Additive number of ibuprofen taken over monitoring period
Number of Tylenol administered | Baseline to 48 hours
  Additive number of acetaminophen taken over monitoring period

SECONDARY OUTCOMES:
Arch Response | Baseline to 48 hours
  Difference in pain response based upon arch
Number of teeth | Baseline to 48 hours
  Difference in pain response based upon number of teeth per surgical site
Type of procedure | Baseline to 48 hours
  Difference in pain response based upon type of procedure
Gender of patient | Baseline to 48 hours
  Difference in pain response based upon gender of participant
Age of patient | Baseline to 48 hours
  Difference in pain response based upon age of participant

CONTACTS AND LOCATIONS:
Overall Officials: David Deas, DDS, MS, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- The University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The PI will share all collected deidentified IPD, all deidentified IPD that underlie results in a publication with colleagues.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared at the time of publication in a peer reviewed journal after the study has completed.